CLINICAL TRIAL: NCT03172104
Title: Neurobehavioural Development of Infants Born <30 Weeks Gestational Age and Their Parents Psychological Wellbeing Between Birth and Five Years of Age
Brief Title: Neurobehavioural Development of Infants Born <30 Weeks Gestational Age Between Birth and Five Years of Age
Acronym: VIBeS-2
Status: Completed | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Principal Investigator, Alicia Spittle, Associate Professor Alicia Spittle, Murdoch Childrens Research Institute
Other Study IDs: HREC34147E
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Preterm Infant; Motor Activity; Neurodevelopmental Disorders; Developmental Coordination Disorder
MeSH Terms: conditions — Premature Birth; Motor Activity; Neurodevelopmental Disorders; Motor Skills Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Very preterm group: Preterm infants <30 weeks' GA at birth admitted to one of the neonatal nurseries at the Royal Women's Hospital in Melbourne, Australia.
  Inclusion criteria: Infants admitted to the Royal Women's Hospital, Melbourne, Australia, neonatal nurseries, born <30 weeks' GA. Exclusion criteria: (i) infants with congenital abnormalities known to affect neurodevelopment and (ii) infants with non-English speaking parents.
- Term control group: Inclusion criteria: Infants admitted to the Royal Women's Hospital Melbourne, Australia, born >36 completed weeks' GA and weighing >2500 g. Exclusion criteria: (i) infants with congenital abnormalities known to affect neurodevelopment (ii) infants requiring admission to neonatal intensive or special care nursery and (iii) infants with non-English speaking parents.

SUMMARY:
Research question: The primary aim of this study is to compare the prevalence of motor impairment from birth to five years of age between children born <30 weeks and term-born controls, and to determine whether persistent abnormal motor assessments in the newborn period in those born <30 weeks predict abnormal motor functioning at age five years. Secondary aims for both children born<30 weeks and term children are i) to determine whether novel early magnetic resonance imaging (MRI) - based structural or functional biomarkers are detectable in the neonatal period that can predict motor impairments at five years, ii) to investigate the association between motor impairments and concurrent deficits in body structure and function at five years of age, and iii) to explore how motor impairments at five years, including abnormalities of gait, postural control and strength, are associated with concurrent functional outcomes including physical activity, cognitive and learning ability, behavioural and emotional problems.

Design: Prospective longitudinal cohort study. Participants and Setting: 150 preterm children (born <30 weeks) and 151 term-born children (born >36 completed weeks' gestation and weighing>2499 g) admitted to the Royal Women's Hospital, Melbourne, were recruited at birth and will be invited to participate in a five-year follow-up study.

Procedure: This study will examine previously collected data (from birth to two years) that comprises the following: detailed motor assessments and structural and functional brain MRI images. At five years, preterm and term children will be examined using comprehensive motor assessments including the Movement Assessment Battery for Children - 2nd edition and measures of gait function through spatiotemporal (assessed with the GAITRite® Walkway), dynamic postural control (assessed with Microsoft Kinect) variables and hand grip strength (assessed with a dynamometer); and measures of physical activity (assessed using accelerometry), cognitive development (assessed with Wechsler Preschool and Primary Scale of Intelligence) and emotional and behavioural status (assessed with the Strengths and Difficulties Questionnaire and the Developmental and Wellbeing Assessment). Caregivers will be asked to complete questionnaires on demographics, physical activity, activities of daily living and motor function (assessed with Pediatric Evaluation of Disability Inventory, Pediatric Quality of Life Questionnaire, the Little Developmental Co-ordination Questionnaire and an activity diary) at the 5 year assessment.

Analysis: For the primary aim the prevalence of motor impairment from birth to 5 years will be compared between children born <30 weeks and term-born peers using the proportion of children classified as abnormal at each of the time points (term age, one, two and five years). Persistent motor impairments during the neonatal period will be assessed as a predictor of severity of motor impairment at 5 years of age in children born <30 weeks using linear regression. Models will be fitted using generalised estimating equations with results reported using robust standard errors, to allow for the clustering of multiple births.

Discussion/Significance: Understanding the developmental precursors of motor impairment in children born <30 weeks is essential to limit disruption to skill development, and potential secondary impacts on physical activity, participation, academic achievement, self-esteem and associated outcomes, such as obesity, poor physical fitness and social isolation. Better understanding of motor skill development will enable targeting of intervention and streamlining of services to the individuals who are at highest risk of motor impairments.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the Royal Women's Hospital, Melbourne, Australia, neonatal nurseries, born <30 weeks' gestational age

Exclusion Criteria:

* (i) infants with congenital abnormalities known to affect neurodevelopment and (ii) infants with non-English speaking parents.

Ages: 0 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants <30 weeks' GA at birth admitted to one of the neonatal nurseries at the Royal Women's Hospital in Melbourne, Australia.
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Motor development | 4.5-5 years corrected age
  Movement Assessment Battery for Children - 2nd Edition

SECONDARY OUTCOMES:
Physical Activity | 4.5-5 years corrected age
  A small Axivity AX3 tri-axial accelerometer-based activity monitor will be worn on the ankle over a consecutive seven day period to obtain information about the number of steps taken per day and sedentary behaviour patterns. The child and caregiver will be educated on wearing the device, and the child will wear it 24 hours a day for seven days before returning it in a pre-paid envelope.
Pediatric Evaluation of Disability Inventory | 4.5-5 years corrected age
  The PEDI-CAT (Pediatric Evaluation of Disability Inventory)25 is a questionnaire that will be used to assess abilities in three functional domains: Daily Activities (e.g. dressing, feeding), Mobility (e.g. transfers, steps and inclines, running and playing) and Social/Cognitive (e.g. interaction, communication, self-management). It provides standard and scaled scores based on normative and disability samples, and is validated for children with a range of physical and behavioural conditions, including children who use mobility devices. Caregivers will complete the PEDI-CAT on an iPad during their child's assessment.
Little DCD Questionnaire | 4.5-5 years corrected age
  The Little Developmental Coordination Disorder Questionnaire (Little DCD)27 is a parent-completed measure which is designed to identify subtle motor problems in children. This questionnaire has been revised to be appropriate for use by parents of children aged five to seven years of age and its concurrent validity has been established with the MABC-2.28
General Cognitive Function | 4.5-5 years corrected age
  General cognitive function will be assessed using the Wechsler Preschool and Primary Scale of Intelligence (Fourth Edition, Australian and New Zealand Standardised Edition; WPPSI-IV).29 The WPPSI-IV has Australasian norms and is the gold standard measure for assessing general intellectual ability. It provides measures of key cognitive domains: full-scale IQ, verbal comprehension, visual-spatial reasoning, fluid reasoning, working memory, and processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Alici J Spittle, PhD, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Murdoch Childrens Research Institute, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spittle AJ, Thompson DK, Brown NC, Treyvaud K, Cheong JL, Lee KJ, Pace CC, Olsen J, Allinson LG, Morgan AT, Seal M, Eeles A, Judd F, Doyle LW, Anderson PJ. Neurobehaviour between birth and 40 weeks' gestation in infants born <30 weeks' gestation and parental psychological wellbeing: predictors of brain development and child outcomes. BMC Pediatr. 2014 Apr 24;14:111. doi: 10.1186/1471-2431-14-111. PMID 24758605
- [Background] Spittle AJ, McGinley JL, Thompson D, Clark R, FitzGerald TL, Mentiplay BF, Lee KJ, Olsen JE, Burnett A, Treyvaud K, Josev E, Alexander B, Kelly CE, Doyle LW, Anderson PJ, Cheong JL. Motor trajectories from birth to 5 years of children born at less than 30 weeks' gestation: early predictors and functional implications. Protocol for a prospective cohort study. J Physiother. 2016 Oct;62(4):222-3. doi: 10.1016/j.jphys.2016.07.002. Epub 2016 Aug 5. PMID 27634166